CLINICAL TRIAL: NCT05269810
Title: Multicenter Double-blinded Randomized Phase 2a Clinical Trial to Evaluate the Efficacy of SA001 for Dry Eye and Mouth Dryness in the Patients With Primary Sjögren's Syndrome
Brief Title: Clinical Study to Investigate the Efficacy of Orally Administered SA001 in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SA001_04
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Primary Sjögren's Syndrome (pSS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): SA001 Low dose
  Interventions: Drug: SA001 Low dose
- Group 2 (Experimental): SA001 Mid dose
  Interventions: Drug: SA001 Mid dose
- Group 3 (Experimental): SA001 High dose
  Interventions: Drug: SA001 High dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SA001 Low dose — 3 tablets b.i.d for 8 weeks
  Arms: Group 1
Drug: SA001 Mid dose — 3 tablets b.i.d for 8 weeks
  Arms: Group 2
Drug: SA001 High dose — 3 tablets b.i.d for 8 weeks
  Arms: Group 3
Drug: Placebo — 3 tablets b.i.d for 8 weeks
  Arms: Placebo

SUMMARY:
This is a phase2a, multicenter, double-blind, placebo control, randomized study to investigate the efficacy and safety of SA001 in subjects with pSS. A total of 28 subjects (including dropout rate of 30%) will be randomized in a 1:1:1:1 ratio to receive 3 different doses of SA001 or placebo everyday for 8 weeks.

Screening visit will be performed within 1 to 2 weeks(run-in period) prior to dosing after signing the informed consent form (ICF). During the run-in period, if necessary, subjects will apply artificial tears in the symptomatic eyes according to the dosage of artificial tears. Only subjects who have completed the run-in period and who are determined to be suitable for the study eligibility(inclusion/exclusion) criteria as a result of the screening evaluations are randomized to one of the four groups.

Subjects will receive investigational product start on Day 0 for 8 weeks during the active treatment period. Subjects will visit to the study site on 4 and 8 weeks after starting dosing investigational product.

Subjects will be in this study approximately 12weeks, which includes run-in period of 1 to 2weeks and a safety follow-up period of 2weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 through 80 years
* Patient who diagnosed with Primary Sjögren's Syndrome(has a score of ≥ 4 when the weights from 5 criteria items are summed) ① Labial salivary gland with focal lymphocytic sialadenitis and focus score of ≥ 1 foci/4 mm2 (weight: 3)

  ② Anti-SSA/Ro-positive (weight: 3)

  ③ Ocular Staining Score ≥ 5 (or van Bijsterveld score ≥ 4) in at least one eye (weight: 1)

  ④ Schirmer's test ≤ 5 mm/5 min in at least one eye (weight: 1)

  ⑤ Unstimulated whole saliva flow rate ≤ 0.1 mL/min (weight: 1)
* Standard Patient Evaluation of Eye Dryness(SPEED) score ≥ 5

Exclusion Criteria:

* Secondary Sjögren's Syndrome patient
* Severe blepharitis caused by Meibomian gland dysfunction
* Administration of eye drops that may affect efficacy assessment in the past 2 weeks prior to baseline (Steroid, glaucoma, allergy, antibiotic, eye drop gel, Cyclosporine, Diquafosol tetrasodium, etc)
* New administration or changing the dosage of systemic steroid drugs or immunosuppressant that may affect immune function in the past 4 weeks prior to baseline
* Administration of oral medication of Tetracycline, Isotretinoin in the past 4 weeks prior to baseline
* New administration or changing the dosage of Hydroxychloroquine medication in the past 12 weeks prior to baseline
* Planning to undergo eye surgery(including eyesight correction surgery) during the study period
* Wearing contact lenses during the study period
* History of ophthalmic surgery and trauma in the past 6 months prior to signing the ICF
* Participation in an investigational drug or device trial within 3 months prior to signing the ICF
* Hypersensitivity to the ingredients of this drug
* Genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* A woman who has a positive Serum hCG test at the screening visit (Visit 1), or who does not agree to use at least one effective contraceptive method that is medically acceptable
* Take oral contraceptives during the study period
* Pregnant or lactating women
* A history of drug or alcohol abuse
* Any condition that, in the opinion of the investigator, would inappropriate to participate in the clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Change in Tear Break-Up Time(TBUT) from baseline to Day 28 and Day 56 | Baseline(Day0), Day 28 and Day 56
Change in Ocular Staining Score(OSS) from baseline to Day 28 and Day 56 | Baseline(Day0), Day 28 and Day 56
Change in Schirmer Test score from baseline to Day 28 and Day 56 | Baseline(Day0), Day 28 and Day 56
Change in Standard Patient Evaluation of Eye Dryness questionnaire(SPEED) score from baseline to Day 28 and Day 56 | Baseline(Day0), Day 28 and Day 56
Change in Unstimulated whole saliva flow rate from baseline to Day 56 | Baseline(Day0) and Day 56
Change in The Xerostomia Inventory(XI) score from baseline to Day 56 | Baseline(Day0) and Day 56
Change in Anti-SSA/Ro levels from baseline to Day 56 | Baseline(Day0) and Day 56
Change in the average number of daily use of the artificial tears from baseline to Day 28 and Day 56 | Baseline(Day0), Day 28 and Day 56
  Artificial tears may be applied if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Yul Seo, Ph.D., Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea